CLINICAL TRIAL: NCT07122986
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, THIRD-PARTY-UNBLINDED STUDY TO EVALUATE THE SAFETY AND TOLERABILITY OF A VACCINE AGAINST E COLI IN HEALTHY ADULTS
Brief Title: A Study to Learn About a Vaccine Against E Coli in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C5211001
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- E coli vaccine 1 Dose A (Experimental): Candidate E coli vaccine on day 1 and day 180
  Interventions: Drug: E coli vaccine 1 Dose A
- E coli vaccine 1 Dose B (Experimental): Candidate E coli vaccine on day 1 and day 180
  Interventions: Drug: E coli vaccine 1 Dose B
- E coli vaccine 2 (Experimental): Candidate E coli vaccine on day 1 and day 180
  Interventions: Drug: E coli vaccine 2
- E coli vaccine 3 (Experimental): Candidate E coli vaccine on day 1 and day 180
  Interventions: Drug: E coli vaccine 3
- E coli Vaccine 4 Dose A (Experimental): Candidate E coli vaccine on day 1 and day 180
  Interventions: Drug: E coli Vaccine 4 Dose A
- E coli Vaccine 4 Dose B (Experimental): Candidate E coli vaccine on day 1 and day 180
  Interventions: Drug: E coli Vaccine 4 Dose B
- E coli Vaccine 4 Dose C (Experimental): Candidate E coli vaccine on day 1 and day 180
  Interventions: Drug: E coli Vaccine 4 Dose C
- E coli Vaccine 5 Dose A (Experimental)
  Interventions: Drug: E coli Vaccine 5 Dose A
- E coli Vaccine 5 Dose B (Experimental)
  Interventions: Drug: E coli Vaccine 5 Dose B
- Placebo (Experimental): Placebo received on day 1 and day 180
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E coli vaccine 1 Dose A — Candidate E coli vaccine 1 Dose A, administered according to a 0, 6-month interval
  Arms: E coli vaccine 1 Dose A
Drug: E coli vaccine 1 Dose B — Candidate E coli vaccine 1 Dose B, administered according to a 0, 6-month interval
  Arms: E coli vaccine 1 Dose B
Drug: E coli vaccine 2 — Candidate E coli vaccine 2, administered according to a 0, 6-month interval
  Arms: E coli vaccine 2
Drug: E coli vaccine 3 — Candidate E coli vaccine 3, administered according to a 0, 6-month interval
  Arms: E coli vaccine 3
Drug: E coli Vaccine 4 Dose A — Candidate E coli vaccine 4 Dose A, administered according to a 0, 6-month interval
  Arms: E coli Vaccine 4 Dose A
Drug: E coli Vaccine 4 Dose B — Candidate E coli vaccine 4 Dose B, administered according to a 0, 6-month interval
  Arms: E coli Vaccine 4 Dose B
Drug: E coli Vaccine 4 Dose C — Candidate E coli vaccine 4 Dose C, administered according to a 0, 6-month interval
  Arms: E coli Vaccine 4 Dose C
Drug: E coli Vaccine 5 Dose A — Candidate E coli vaccine 5 Dose A, administered according to a 0, 6-month interval
  Arms: E coli Vaccine 5 Dose A
Drug: E coli Vaccine 5 Dose B — Candidate E coli vaccine 5 Dose B, administered according to a 0, 6-month interval
  Arms: E coli Vaccine 5 Dose B
Drug: Placebo — Placebo administered according to a 0, 6-month interval
  Arms: Placebo

SUMMARY:
This study evaluates an investigational vaccine designed to protect against Escherichia coli (E coli). The primary objective is to assess the safety and tolerability of E coli vaccines administered intramuscularly to healthy adults.

ELIGIBILITY:
Ages Eligible for Study: 18 to 64 Years (Adult) Sexes Eligible for Study: All Accepts Healthy Volunteers: Yes

Key Inclusion Criteria

1. Adult Participants >= 18 through < 64 years of age at the time of enrollment.
2. Healthy participants as determined by medical history, physical examination, and clinical judgement of the investigator to be eligible for inclusion in the study.

Key Exclusion Criteria

1. Severe adverse reaction history associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
2. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
3. Women who are pregnant, plan to become pregnant during the study, or are breastfeeding.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2028-05-26 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting prespecified local events within 7 days following each vaccination | 7 days after each vaccination
  Prespecified local reactions (redness, swelling, and pain at the injection site) following each vaccination
Percentage of participants reporting prespecified systemic events within 7 days following each vaccination | 7 days after each vaccination
  Prespecified systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, joint pain, and muscle pain) following each vaccination
Percentage of participants reporting Adverse Events (AEs) from vaccination 1 through 1 month after the last dose of study intervention | From signing of ICD to 1 month after the last assigned vaccination
  Adverse events occurring up to 1 month after the last dose of study intervention
Percentage of participants reporting Medically Attended Adverse Events (MAEs) from vaccination 1 through 12 months after the last dose of study intervention | Baseline up to month 18 with final visit being 12 months after last assigned vaccination
  MAEs occurring up to 12 months after the last dose of study intervention
Percentage of participants reporting Serious Adverse Events (SAEs) from vaccination 1 through 12 months after the last dose of study intervention | Baseline up to month 18 with final visit being 12 months after last assigned vaccination
  SAEs occurring up to 12 months after the last dose of study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Orange County Research Center, Lake Forest, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Miami Eye Institute, Hollywood, Florida
  - Research Centers of America, Hollywood, Florida
  - NYU Langone Health, New York, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - University Eye Specialists, P.C. (Ophthalmologist), Maryville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5211001